CLINICAL TRIAL: NCT03661931
Title: Dietary Quality Photo Navigation: A Preliminary Biomarker Validation Study and Comparison With a Food Frequency Questionnaire
Brief Title: Dietary Quality Photo Navigation (DQPN) Preliminary Validation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Boston Heart Diagnostics (Industry)
Collaborators: David M. Katz, M.D. (Individual)
Responsible Party: Principal Investigator, Michael Dansinger, Principal Investigator, Boston Heart Diagnostics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BHD-005
Record Dates: First submitted 2018-09-04; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Lifestyle-related Condition; Nutrient; Excess
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DQPN Validation (Experimental): We are planning to recruit 150 individuals who are patients in the Boston Heart Lifestyle Program and are already having fatty acids measured as part of clinical care, and ask them to complete the DQPN, FFQ, and a User Experience Questionnaire for each dietary assessment method.
  Interventions: Diagnostic Test: DQPN Validation

INTERVENTIONS:
Diagnostic Test: DQPN Validation — We are planning to recruit 150 individuals who are patients in the Boston Heart Lifestyle Program and are already having fatty acids measured as part of clinical care, and ask them to complete the DQPN, FFQ, and a brief User Experience Questionnaire for each dietary assessment method.

SUMMARY:
The purpose of this research project is to conduct a preliminary validation study of the Diet Quality Photo Navigation (DQPN) method of dietary intake assessment. In 150 adults, dietary intake as estimated by the DQPN will be compared to dietary intake as estimated by a food frequency questionnaire (FFQ) and with blood levels of fatty acids, folic acid, and beta-carotene as biomarkers of dietary intake.

DETAILED DESCRIPTION:
The primary aim is to test thee principal hypotheses (n=150):

1. There will be statistically significant correlations between blood levels of fatty acids/folate/beta-carotene and their corresponding levels of dietary intake as estimated by the DQPN.
2. There will be statistically significant correlations between the DQPN and FFQ methods of dietary intake assessment. This includes individual dietary components as well as overall dietary quality and disease risk assessments.
3. User experience surveys will demonstrate that the DQPN can be completed more quickly and more enjoyably than the FFQ.

In addition, investigators will assess whether blood levels of fatty acids/folate/beta-carotene are similarly associated with the DQPN method and the FFQ method, and will measure the test-retest reliability of the DQPN method.

ELIGIBILITY:
Inclusion Criteria:

* Clinical provider has ordered fasting Boston Heart Fatty Acid Balance and participation in the Boston Heart Lifestyle Program as part of clinical practice.
* Willing to fill out Food Frequency Questionnaire
* Willing to complete DQPN Diet IDTM (on-line), and to repeat that 1 week later
* Willing to complete user experience surveys about each dietary assessment method

Exclusion Criteria:

* Taking fatty acid or vitamin supplements (such as fish oil capsules, or multivitamin tablets)
* Following a diet outside the capabilities of the DQPN cannot be included in this study. The vast majority of eating styles are within the assessment capabilities of the DQPN (Standard American, Low-fat, Mediterranean, Pescatarian, Flexitarian, Low-carb, DASH, AHA, TLC, MIND, Vegetarian, Vegan, Paleo, Southern).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-11 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between DQPN results and FFQ results | 6 months
  The primary outcome is the set of correlation coefficients comparing the DQPN results and the FFQ results

SECONDARY OUTCOMES:
Correlation between DQPN and biomarkers | 6 months
  A secondary outcome is the set of correlation coefficients comparing the DQPN results and the corresponding blood levels of fatty acids, folic acid, and beta-carotene
Number of minutes spent completing the DQPN and FFQ | 6 months
  A secondary outcome is the median number of minutes spent completing the DQPN and the FFQ will be compared
Correlation between FFQ and biomarkers | 6 months
  A secondary outcome is the set of correlation coefficients comparing the FFQ results and the corresponding blood levels of fatty acids, folic acid, and beta-carotene.
Retest reliability for DQPN | 6 months
  A secondary outcome is the test-retest reliability coefficient (tau-equivalent reliability measurement) for the DQPN

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dansinger, MD, Principal Investigator — Boston Heart Diagnostics

IPD SHARING:
Plan to Share IPD: No